CLINICAL TRIAL: NCT04906850
Title: Comparison of Mortality in Severe SARS-Cov-2 Infection Caused by the 501Y.V2 Variant and B.1.1.7 Variant
Brief Title: Evaluation of the New Variant 501Y.V2 of COVID-19
Acronym: VARICOVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-05Obs-CHRMT
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: Mortality; SARS-CoV-2 variants; Intensive Care Unit; 20I/501Y.V1; 20H/501Y.V2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In January 2021, the incidence of COVID-19-and its mortality started rising for the third time in France. This rise may associate with three emerging variants, namely, V1, V2, and V3, which are the 20I/501Y.V1 ("English"), 20H/501Y.V2 ("South African"), and 20J/501Y.V3 ("Brazilian") variants, respectively. V1 was recently suggested to increase mortality in people in the United Kingdom who tested positive for COVID-19 on community screening. Very little is known about V2 infection, including its outcomes relative to other strains. In early 2021, V2 spread to the Grand-Est region (northeastern France). Here, the investigators aimed to report mortality data of patients admitted in ICU between February and April 2021 in 3 hospitals in Grand-Est: Metz, Thionville and Nancy.

ELIGIBILITY:
Inclusion Criteria:

* Admission in ICU in February, March or April 2021
* Patient with a SARS-CoV-2 positive polymerase-chain reaction test
* Patient with 20I/501Y.V1 ("English") or 20H/501Y.V2 ("South African") SARS-CoV-2 variants

Exclusion Criteria:

* Opposed to use data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with 20I/501Y.V1 ("English") or 20H/501Y.V2 ("South African") SARS-CoV-2 variants
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Mortality 28 days after admission | Day 28
  Vital status 28 days after admission in Intensive Care Unit

SECONDARY OUTCOMES:
ICU mortality | Day 1
  Percentage of mortality in Intensive Care Unit

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU Nancy, Nancy, Meurthe-et-moselle
  - CHR Metz Thionville, Metz, Moselle

REFERENCES:
- [Derived] Louis G, Belveyre T, Goetz C, Gibot S, Dunand P, Conrad M, Gaci R, Gette S, Ouamara N, Perez P, Cadoz C, Picard Y, Mellati N. Comparison of SARS-CoV-2 Variants of Concern Alpha (B.1.1.7) vs. Beta (B.1.351) in Critically Ill Patients: A Multicenter Cohort Study. Front Med (Lausanne). 2022 Mar 10;9:828402. doi: 10.3389/fmed.2022.828402. eCollection 2022. PMID 35360736